CLINICAL TRIAL: NCT07039370
Title: The Relationship Between Plasma Metabolomics and Proteomics Profiling and Response to Transcranial Magnetic Stimulation Therapy in Treatment-Resistant Depression
Brief Title: Molecular Signatures of TMS Response in Treatment-Resistant Depression
Acronym: PROMET_TMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Beyazit Garip, Principal Investigator, Gulhane Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025/245 / 46418926
Record Dates: First submitted 2025-05-31; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Major Depression Disorder
Keywords: TMS; Metabolomics; Proteomics; Treatment Resistance; Molecular Signuture

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-group, open-label cohort study designed to evaluate the association between plasma proteomic and metabolomic profiles and clinical response to transcranial magnetic stimulation (TMS) in patients with treatment-resistant depression (TRD). All participants in the intervention arm will receive a standardized TMS protocol targeting the left dorsolateral prefrontal cortex. A group of age- and sex-matched healthy individuals will serve as a non-randomized control group for baseline biomarker comparison. No randomization or blinding will be employed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcranial Magnetic Stimualtion Treatment Arm (Experimental): This arm includes participants diagnosed with treatment-resistant depression (TRD) who will receive transcranial magnetic stimulation (TMS) therapy. TMS will be delivered using the MagVenture™ X100™ device. The treatment protocol consists of 20 sessions over a 4-week period (5 sessions per week). Stimulation will target the left dorsolateral prefrontal cortex (DLPFC) using intermittent theta burst stimulation (iTBS). Motor threshold will be determined at baseline and reassessed weekly to calibrate stimulation intensity at 90% of the resting motor threshold.
  Blood samples will be collected from participants at two time points: prior to the first TMS session (pre-treatment) and following the final (20th) session (post-treatment). Proteomic and metabolomic analyses will be performed using high-resolution liquid chromatography-mass spectrometry (LC-MS). The goal is to identify differentially expressed proteins and metabolites associated with clinical response to TMS.
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — Transcranial Magnetic Stimulation (TMS) is a non-invasive brain stimulation technique approved for the treatment of major depressive disorder (MDD), particularly in individuals with treatment-resistant depression (TRD). TMS targets the left dorsolateral prefrontal cortex (DLPFC), a brain region often underactive in depression, and modulates neural activity through magnetic pulses.
  This study aims to evaluate the effects of TMS on plasma proteomic and metabolomic profiles in patients with TRD. Participants will undergo 20 sessions of intermittent theta burst stimulation (iTBS) over four weeks. Blood samples will be collected before and after treatment to identify molecular changes associated with clinical response. Healthy controls will provide single-time-point blood samples for baseline comparison. Findings may support the development of biomarker-based strategies for personalized treatment in psychiatry.

SUMMARY:
Transcranial Magnetic Stimulation (TMS) therapy is an approved and effective treatment option for treatment-resistant depression (TRD). This study aims to identify biomarkers that predict TMS treatment response in TRD, provide insights into the neurobiological mechanisms underlying TMS efficacy, and contribute to personalized treatment strategies. By establishing proteomic and metabolomic signatures, this research seeks to enhance clinical decision-making, reduce healthcare costs, and improve patient outcomes in TRD. The findings will align with the precision medicine movement in psychiatry, advancing biomarker-driven therapeutic approaches for treatment-resistant depression.

DETAILED DESCRIPTION:
This prospective cohort study aims to investigate the relationship between plasma proteomic and metabolomic profiles and the treatment response to transcranial magnetic stimulation (TMS) in patients with treatment-resistant depression (TRD). TRD is defined as a subtype of major depressive disorder (MDD), characterized by an inadequate response to at least two adequate trials of antidepressant therapy. Despite the clinical efficacy of TMS as a non-invasive neuromodulation treatment, the biological underpinnings that determine patient responsiveness remain unclear. This study addresses that gap by evaluating blood-based molecular biomarkers that may predict or reflect TMS treatment outcomes.

A total of 55 TRD patients, diagnosed according to DSM-5-TR criteria and confirmed through the SCID-5 structured clinical interview, will be enrolled. An additional 55 healthy individuals matched for age and sex will serve as a control group for baseline plasma comparisons. Patients will undergo a standardized TMS protocol using the MagVenture™ X100™ device. The protocol includes 20 treatment sessions over four weeks, with each session delivering 1,800 pulses of intermittent theta burst stimulation (iTBS) targeting the left dorsolateral prefrontal cortex (DLPFC). Motor threshold will be assessed weekly to calibrate treatment intensity to 90% of the resting motor threshold.

Blood samples will be collected from TRD patients prior to the first TMS session and after the 20th session, while healthy controls will provide samples at a single time point. Proteomic analysis will be conducted using LC-MS/MS following protein extraction, digestion, and purification. Metabolomic profiling will be carried out using LC-MS coupled with ion mobility spectrometry, enabling the identification of a wide range of plasma metabolites.

Psychiatric assessments, including the Hamilton Depression Rating Scale (HAM-D), Patient Health Questionnaire-9 (PHQ-9), Pittsburgh Sleep Quality Index (PSQI), and the Clinical Global Impression (CGI) scale, will be administered at baseline and post-treatment to monitor clinical outcomes. Data integration and bioinformatics analyses will be performed using MaxQuant, Perseus, and MetaboAnalyst 6.0, enabling the identification of differentially expressed proteins and metabolites associated with treatment response.

The primary objective of the study is to determine whether plasma proteomic and metabolomic profiles differ significantly between TMS responders and non-responders. Secondary objectives include identifying predictive biomarkers for TMS efficacy and assessing biological changes correlated with clinical improvement.

Primary outcomes will focus on identifying molecular signatures that correlate with treatment responsiveness. Secondary outcomes will include changes in depression severity scores, documentation of any adverse effects related to TMS, and examination of correlations between biomarker expression and pharmacological history.

This study is crucial for advancing personalized treatment approaches in psychiatry. By identifying objective, blood-based biomarkers of TMS response, it may become possible to tailor treatment strategies, reduce unnecessary interventions, and improve therapeutic outcomes for individuals suffering from TRD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder (MDD) according to DSM-5-TR criteria.
* Inadequate clinical response to at least two different antidepressants and/or anti-obsessive agents administered at therapeutic doses and durations.
* Clinical symptoms not better explained by metabolic or organic medical conditions.
* No epileptic activity detected on routine electroencephalography (EEG) prior to TMS initiation.
* Routine pre-TMS laboratory tests reveal no abnormalities that may significantly affect treatment response, including:
* Normal thyroid hormone profile
* No significant vitamin deficiencies
* No markedly elevated inflammatory markers
* No history or current evidence of hearing loss on clinical evaluation; if present, evaluation by an otolaryngologist will be obtained.
* Age 18 years and older.
* Ability to provide written informed consent.

Exclusion Criteria:

* Any contraindication to TMS as identified in the standardized pre-TMS risk assessment form.
* Presence of epileptic focus detected on pre-TMS EEG.
* History of significant head trauma, loss of consciousness, or intracranial surgery.
* Presence of metal implants or foreign bodies incompatible with TMS (e.g., aneurysm clips, surgical clamps, metallic fragments).
* Abnormal thyroid hormone levels in pre-TMS laboratory testing.
* Significantly elevated inflammation markers (e.g., CRP) in pre-TMS bloodwork.
* Vitamin deficiencies associated with cognitive impairment (e.g., B12, folate) in pre-TMS labs.
* Electrolyte imbalances on pre-TMS blood testing.
* History of psychotic disorder or bipolar I/II disorder.
* History of substance-induced psychosis or bipolar disorder.
* Current or past substance use disorder (including alcohol, stimulants, or illicit drugs), unless abstinent from substances (excluding alcohol) for a minimum of 12 months.
* Voluntary discontinuation of TMS during the treatment course.
* Any serious adverse event or unexpected clinical condition during treatment that necessitates discontinuation of TMS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Plasma Proteomic Profile Changes After TMS in Patients with Treatment-Resistant Depression | From enrollment to end of treatment at 4 weeks
  Assessment of differences in plasma proteomic profiles in treatment-resistant depression (TRD) patients before and after transcranial magnetic stimulation (TMS), using high-resolution liquid chromatography-mass spectrometry (LC-MS/MS) analysis. Changes in protein expression will be used to identify potential biomarkers of treatment response.
Plasma Metabolomic Profile Changes After TMS in Patients with Treatment-Resistant Depression | From enrollment to end of treatment at 4 weeks
  Evaluation of global metabolomic changes in plasma of TRD patients pre- and post-TMS therapy. Analysis will be conducted via liquid chromatography-mass spectrometry with ion mobility separation (LC-TIMS-TOF-MS), enabling identification of differential metabolites associated with clinical outcomes.
Fold Change in Baseline Proteomic Markers Between Treatment Responders and Non-Responders | From enrollment to end of the treatment at 4 weeks
  Differences in baseline proteomic markers between treatment responders and non-responders will be assessed using LC-MS/MS. Fold change values will be calculated to identify proteins with significant differential expression between the two groups.
Variable Importance in Projection Scores of Predictive Proteins | Baseline and End of 4-week treatment
  Variable Importance in Projection scores will be calculated using multivariate statistical analysis (e.g., PLS-DA) to rank the importance of baseline proteomic markers in distinguishing treatment responders from non-responders.
Area Under the ROC Curve for Predictive Proteomic Markers Between Treatment Responders and Non-Responders | Baseline and End of 4-week treatment
  Receiver Operating Characteristic (ROC) curve analysis will be performed to evaluate the predictive performance of baseline and end-of-treatment proteomic markers in distinguishing treatment responders from non-responders. Area Under the Curve (AUC) values will be calculated to assess discriminative ability.
Fold Change in Baseline Plasma Metabolomic Markers Between TMS Responders and Non-Responders | Baseline
  Fold change in baseline plasma metabolomic expression levels will be assessed between TMS treatment responders and non-responders using LC-MS/MS. The analysis aims to identify significantly altered metabolites that may predict treatment response.
Variable Importance in Projection Scores of Baseline Plasma Metabolomic Markers Between TMS Responders and Non-Responders | Baseline and End of 4-week treatment
  Variable Importance in Projection scores will be calculated using multivariate statistical models (e.g., PLS-DA) to rank baseline plasma metabolomic markers according to their importance in differentiating TMS treatment responders from non-responders.
  Unitless
Area Under the ROC Curve of Baseline Plasma Metabolomic Markers Between TMS Responders and Non-Responders | Baseline and End of 4-week treatment
  Receiver Operating Characteristic curve analysis will be conducted to evaluate the predictive accuracy of baseline plasma metabolomic markers in distinguishing TMS treatment responders from non-responders. The Area Under Curve (AUC)will quantify each marker's discriminative ability. Measurement Tool:
  ROC curve analysis
  Unit of Measure: AUC (0-1 scale)

SECONDARY OUTCOMES:
Change in Depression Severity Based on Hamilton Depression Rating Scale (HAM-D, 17-item) | From enrollment to the end of the treatment at 4 weeks
  Depression severity will be assessed using the 17-item clinician-administered HAM-D scale. Scores range from 0 to 34, with higher scores indicating more severe depressive symptoms. A clinical response is defined as a ≥50% reduction in HAM-D total score from baseline to post-treatment
Change in Depression Severity Based on Patient Health Questionnaire-9 (PHQ-9) | From enrollment to the end of the treatment at 4 weeks
  Depression severity will be self-assessed by participants using the PHQ-9 scale. Scores range from 0 to 27, with higher scores reflecting more severe symptoms. A clinical response is defined as a ≥50% reduction in PHQ-9 total score from baseline to post-treatment.
Change in Subjective Sleep Quality Measured by Pittsburgh Sleep Quality Index [Sleep Quality] | From enrollment to end of the treatment 4 weeks
  Subjective sleep quality will be assessed using the Pittsburgh Sleep Quality Index(PSQI) a self-reported questionnaire consisting of 24 items that evaluate sleep quality over the past month across seven domains (e.g., sleep latency, duration, disturbances). Total score range: 0 to 21. Minimum possible score: 0 (indicating good sleep quality). Maximum possible score: 21 (indicating poor sleep quality). Interpretation: Higher scores indicate worse sleep quality. Changes in PSQI total scores from baseline to the end of the 4-week treatment period will be analyzed.
Correlation Between Antidepressant Medication Use and Clinical Response to TMS Measured by Hamilton Depression Rating Scale-17 | From enrollment to end of the treatment at 4 weeks
  This outcome will assess the correlation between concurrent antidepressant medication use and clinical response to Transcranial Magnetic Stimulation (TMS). Medication data collected: Drug name, dosage, duration. Clinical outcome: Change in Hamilton Depression Rating Scale-17 (HAM-D17) total score from baseline to end of treatment. Statistical method: Pearson or Spearman correlation (based on data distribution). Unit of Measure (Antidepressant Use): Continuous (daily dose in mg), duration in weeks. Unit of Measure (TMS Response): Change in HAM-D17 total score
Change in Headache and Scalp Pain Severity Measured by Visual Analog Scale (VAS) [Tolerability] | Baseline and End of 4-week treatment
  Change in Headache and Scalp Pain Severity Measured by Visual Analog Scale (VAS) [Tolerability]
Incidence of Seizure Events | From enrollment to end of the 4 weeks
  The number and percentage of participants who experience seizures during the 4-week treatment period will be recorded. Events will be classified according to severity and assessed for their relationship to the study intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IDP) will be shared together with the Clinical Study Report
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be made available immediately after the publication, and will remain available for at least 5 years.
Access Criteria: Anyone who wishes to access the data